CLINICAL TRIAL: NCT02857816
Title: PRospective Study to Evaluate EffectivenesS With the NURO™ PErcutaneous Tibial Neuromodulation (PTNM) System in Patients With OAB
Brief Title: PRospective Study to Evaluate EffectivenesS With the NURO™ PErcutaneous Tibial Neuromodulation System in Patients With OAB
Acronym: RESET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1679
Record Dates: First submitted 2016-08-03; First posted 2016-08-05 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2018-12

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- NURO System PTNM Therapy (Other): Subjects will undergo 12 PTNM therapy sessions, administered weekly, utilizing the NURO system.
  Interventions: Device: NURO System PTNM Therapy

INTERVENTIONS:
Device: NURO System PTNM Therapy

SUMMARY:
To evaluate the NURO system for the treatment of OAB in drug naïve patients.

DETAILED DESCRIPTION:
The purpose of this prospective, multicenter, single arm study is to evaluate the NURO system for the treatment of OAB in drug naïve patients. The study will assess change from baseline through 12 PTNM therapy sessions in UUI (urge urinary incontinence) episodes, voiding episodes, and patient reported outcomes. The study is expected to last approximately 14 weeks per subject following the enrollment visit. Subjects will be exited from the study after the final study visit is complete.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Diagnosis of OAB and associated symptoms of UUI and qualify with at least 3 episodes of mild, moderate, or severe urgency demonstrated on a 3-day urinary voiding diary
3. Experiencing UUI symptoms for at least 3 months
4. No prior treatment with anticholinergics/antimuscarinics or beta 3-agonists medications to treat OAB
5. Willing and able to accurately complete voiding diaries and questionnaires, attend visits, and comply with the study protocol
6. Willing and able to provide signed and dated informed consent

Exclusion Criteria:

1. Have received anticholinergics/antimuscarinics or beta 3-agonists medications to treat OAB or advanced therapy treatment options for OAB (botulinum toxin injections, sacral neuromodulation, or percutaneous tibial nerve stimulation/neuromodulation)
2. Primary stress incontinence or mixed incontinence where the stress component overrides the urge component
3. Have implantable pacemakers or implantable defibrillators
4. Use of transcutaneous electrical nerve stimulation (TENS) in pelvic region, back or legs
5. Women who are pregnant or planning to become pregnant during the course of the study
6. Characteristics indicating a poor understanding of the study or characteristics that indicate the subject may have poor compliance with the study protocol
7. Nerve damage that could impact either tibial nerve or pelvic floor function.
8. Subjects prone to excessive bleeding
9. Inadequate skin integrity in the area of PTNM needle placement
10. History of diabetes unless the diabetes is well-controlled through diet and/or medications
11. Have symptomatic urinary tract infection (UTI)
12. Participation in any research study involving or impacting gynecologic, urinary or renal function within the 4-week period prior to or plans to participate during study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-09; Primary Completion 2017-11-21 (Actual); Study Completion 2017-11-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Pinellas Urology, Inc., St. Petersburg, Florida
  - NorthShore University Health System, Evanston, Illinois
  - Mount Auburn Hospital, Cambridge, Massachusetts
  - Advanced Urogynecology of Michigan, P.C., Dearborn, Michigan
  - Metro Urology, Woodbury, Minnesota
  - Urology Center Research Institute, LLC, Englewood, New Jersey
  - NYU Urology Associates, New York, New York
  - Alliance Urology Specialists, Greensboro, North Carolina
  - Hospital of University of Pennsylvania, Philadelphia, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington
  - SSM Health Dean Medical Group, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred fifty-four subjects were enrolled (consented) to participate in the trial from September 15, 2016 through August 14, 2017 from 12 US centers.
Pre-assignment Details: Out of 154 enrolled subjects, 120 were qualified and 121 subjects received PTNM therapy, with 1 not meeting eligibility criteria.
Groups:
- NURO System PTNM Therapy: Subjects will undergo 12 PTNM therapy sessions, administered weekly, utilizing the NURO system to receive PTNM Therapy
Period: Overall Study
Arm/Group | NURO System PTNM Therapy
Started | 154
Subjects Qualified and Treated With PTNM (This includes those subjects that met eligibility criteria and received PTNM therapy in the study.) | 120
Completed | 116
Not Completed | 38
Not completed — Screen Failure | 33
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: One hundred twenty subjects were qualified for study participation and received PTNM therapy.
Groups:
- NURO System PTNM Therapy: Subjects will undergo 12 PTNM therapy sessions, administered weekly, utilizing the NURO system.
  NURO System PTNM Therapy
Arm/Group | NURO System PTNM Therapy
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 110
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 120
Years since OAB diagnosis [Mean (Standard Deviation); unit: years] | 3.4 (5.1)
Baseline UUI episodes/day [Mean (Standard Deviation); unit: episodes] — Population: One subject did not have evaluable diary data at baseline.
  episodes
    number analyzed (Participants) | 119
    (all) | 3.5 (2.5)
Baseline voids/day [Mean (Standard Deviation); unit: episodes] — Population: Baseline voids/day is only summarized on UF subjects (defined as at least 8 voids/day at baseline). This was not required for study eligibility.
  episodes
    number analyzed (Participants) | 86
    (all) | 11.5 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Urinary Urge Incontinence (UUI) Episodes Per Day After the 12th PTNM Therapy Sessions From Baseline
Description: Number of UUI episodes were collected at baseline and following the 12th PTNM therapy session. For each subject in the analysis, change in UUI episodes per day was calculated as UUI episodes per day after 12th PTNM session minus baseline. A negative change indicates the improvement in UUI symptom.
Time Frame: 12 Weeks
Population: Subjects with diary data from both baseline and the 12th PTNM therapy session
Measure: Mean (Standard Deviation); unit: UUI episodes per day
Arm/Group | NURO System PTNM Therapy
Number analyzed (Participants) | 116
UUI episodes per day | -2.4 (2.1)
Statistical Analysis 1: Comparison: NURO System PTNM Therapy; This is a single arm study. The primary objective was to demonstrate a statistically significant reduction between baseline and following the 12th PTNM therapy sessions in the number of UUI episodes per day; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Number of Voids Per Day After the 12th PTNM Therapy Sessions From Baseline in UF Subjects
Description: Number of voids were collected at baseline and following the 12th PTNM therapy session. For each UF subject in the analysis, a change in number of voids per day was calculated as number of voids per day after 12th PTNM session minus baseline. A negative change indicates improvement in UF symptoms.
Time Frame: 12 Weeks
Population: This objective was assessed in qualified subjects with > 8 voids per day at baseline, who had diary data at both baseline and following the 12th PTNM session.
Measure: Mean (Standard Deviation); unit: Number of voids per day
Arm/Group | NURO System PTNM Therapy
Number analyzed (Participants) | 84
Number of voids per day | -1.7 (2.5)

3. Secondary Outcome: Change in Overactive Bladder Symptom Quality of Life Questionnaire (OABq) After 12th PTNM Therapy Sessions From Baseline
Description: This objective was to assess the change after12 PTNM therapy sessions from baseline in quality of life as measured by the OABq Questionnaire.
  OABq consists of a symptom bother scale and four health related quality of life (HRQL) subscales (Coping, Concern, Sleep and Social interaction). The symptom bother scale and 4 HRQL subscales are measured as 0-100 using a range percentile transformation on the summed value from individual listed items. The HRQL score is a calculated score with a range from 0 to 100 using a range percentile transformation on the summed value from 4 subscales (Coping, Concern, Sleep and Social). A change was calculated as the score after 12th PTNM minus the score at baseline. A positive change in HRQL and its subscales (Coping, Concern, Sleep and Social) indicates improvement in QOL; a negative change in symptom bother score indicates improvement in QOL.
Time Frame: 12 Weeks
Population: This objective was assessed in all qualified subjects who received PTNM therapy and had OABq questionnaire data available at both baseline and 12th PTNM session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NURO System PTNM Therapy
Number analyzed (Participants) | 116
score on a scale
  Concern | 40 (25.8)
  Coping | 32.5 (23.9)
  Sleep | 30.5 (26.9)
  Social | 15.3 (21.8)
  HRQL | 30.7 (20.9)
  Symptom Bother | -43.9 (22.5)

ADVERSE EVENTS:
Time Frame: Adverse events report collected starting from the time of enrollment until completion of the final study visit (approximately 16 weeks).
Description: The following adverse events were considered reportable in accordance with the Clinical Investigational Plan: serious, device related, and/or therapy/procedure related.
Groups:
- NURO System PTNM Therapy: Subjects will undergo 12 PTNM therapy sessions, administered weekly, utilizing the NURO system to receive PTNM Therapy.
  In the summary of serious AEs below, none of the serous AEs were found to be related to device, therapy or study procedure. The other events reported in this study were non-serious device related and/or therapy/procedure related.
Arm/Group | NURO System PTNM Therapy
All-Cause Mortality (participants affected / at risk) | 0/121
Serious Adverse Events (participants affected / at risk) | 3/121
Other Adverse Events (participants affected / at risk) | 8/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NURO System PTNM Therapy (N=121)
Diarrhoea infectious (Infections and infestations) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NURO System PTNM Therapy (N=121)
Medical device site pain (General disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5)

LIMITATIONS AND CAVEATS:
Study had a single arm with all subjects treated with PTNM Therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-06-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT02857816/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT02857816/SAP_001.pdf